CLINICAL TRIAL: NCT00539214
Title: Non-motor Symptoms (Depressive Symptoms) of Parkinson's Disease and Their Course Under Pramipexole Treatment
Brief Title: Non-interventional Observational Study With Pramipexole: Impact on Non-motor Symptoms in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.639
Record Dates: First submitted 2007-09-28; First posted 2007-10-04 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
* To compare the effect of pramipexole on depressive symptoms in early and advanced PD patients
* To evaluate the course of depressive symptoms measured with UPDRS Part I (mentation, behavior and mood) and with HADS-D under pramipexole treatment
* To investigate whether improvement of depressive symptoms is linked to improvement in motor function (UPDRS Part III)

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Idiopathic Parkinsons disease with or without fluctuations
2. Indication for treatment with Sifrol®
3. Male or female patients of age
4. Presence of at least mild depressive symptoms (as judged by the treating physician)
5. Ability to reliably complete a self-rating scale (HADS)

Exclusion criteria:

1. Any contraindications according to the Summary of Product Characteristics (SPC): hypersensitivity to pramipexole or to any of the excipients.
2. Ongoing treatment with Sifrol®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Non-Probability Sample
Enrollment: 1192 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Improvement of depressive symptoms (UPDRS item 3, HADS-D) compared to baseline in early and advanced Parkinsons's disease | 9-16 weeks
Change in sum scores of UPDRS Part III (motor examination) from baseline and UPDRS Part I (mentation, behavior and mood) from baseline | 9-16 weeks
Change in HADS subscores (anxiety and depression) from baseline | 9-16 weeks

SECONDARY OUTCOMES:
Baseline pattern of patient rated symptom list (HADS) | 9-16 weeks
Correlation of the change in UPDRS Part I and UPDRS Part III at the final visit | 9-16 weeks
Frequency of adverse events | 9-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (317):
- Germany (317):
  - Boehringer Ingelheim, Aalen
  - Boehringer Ingelheim, Aarbergen
  - Boehringer Ingelheim, Adendorf
  - Boehringer Ingelheim, Aham
  - Boehringer Ingelheim, Ahaus
  - Boehringer Ingelheim, Ahlen
  - Boehringer Ingelheim, Ahorntal
  - Boehringer Ingelheim, Aichach
  - Boehringer Ingelheim, Aislingen
  - Boehringer Ingelheim, Albstadt
  - Boehringer Ingelheim, Aldenhoven
  - Boehringer Ingelheim, Aldingen
  - Boehringer Ingelheim, Alfeld
  - Boehringer Ingelheim, Alpirsbach
  - Boehringer Ingelheim, Alsdorf
  - Boehringer Ingelheim, Altena
  - Boehringer Ingelheim, Altenstadt
  - Boehringer Ingelheim, Altomünster
  - Boehringer Ingelheim, Alveslohe
  - Boehringer Ingelheim, Amberg
  - Boehringer Ingelheim, Ammerbuch
  - Boehringer Ingelheim, Andernach
  - Boehringer Ingelheim, Anklam
  - Boehringer Ingelheim, Apolda
  - Boehringer Ingelheim, Armsheim
  - Boehringer Ingelheim, Arzberg
  - Boehringer Ingelheim, Aschaffenburg
  - Boehringer Ingelheim, Aschersleben
  - Boehringer Ingelheim, Aschheim
  - Boehringer Ingelheim, Attendorn
  - Boehringer Ingelheim, Auerbach
  - Boehringer Ingelheim, Augsburg
  - Boehringer Ingelheim, Aurich
  - Boehringer Ingelheim, Babensham
  - Boehringer Ingelheim, Backnang
  - Boehringer Ingelheim, Bad Arolsen
  - Boehringer Ingelheim, Bad Berleburg
  - Boehringer Ingelheim, Bad Bevensen
  - Boehringer Ingelheim, Bad Düben
  - Boehringer Ingelheim, Bad Dürrenberg
  - Boehringer Ingelheim, Bad Dürrheim
  - Boehringer Ingelheim, Bad Ems
  - Boehringer Ingelheim, Bad Essen
  - Boehringer Ingelheim, Bad Kreuznach
  - Boehringer Ingelheim, Bad Laasphe
  - Boehringer Ingelheim, Bad Langensalza
  - Boehringer Ingelheim, Bad Lausick
  - Boehringer Ingelheim, Bad Münstereifel
  - Boehringer Ingelheim, Bad Oeynhausen
  - Boehringer Ingelheim, Bad Salzungen
  - Boehringer Ingelheim, Bad Schwalbach
  - Boehringer Ingelheim, Bad Schwartau
  - Boehringer Ingelheim, Bad Segeberg
  - Boehringer Ingelheim, Bad Tennstedt
  - Boehringer Ingelheim, Bad Waldsee
  - Boehringer Ingelheim, Baden-Baden
  - Boehringer Ingelheim, Bahrdorf
  - Boehringer Ingelheim, Baltmannsweiler
  - Boehringer Ingelheim, Bamberg
  - Boehringer Ingelheim, Barleben
  - Boehringer Ingelheim, Baunatal
  - Boehringer Ingelheim, Bautzen
  - Boehringer Ingelheim, Bayreuth
  - Boehringer Ingelheim, Bärnau
  - Boehringer Ingelheim, Beckum
  - Boehringer Ingelheim, Beeskow
  - Boehringer Ingelheim, Bellheim
  - Boehringer Ingelheim, Belm
  - Boehringer Ingelheim, Bensheim
  - Boehringer Ingelheim, Berching
  - Boehringer Ingelheim, Bergfelde
  - Boehringer Ingelheim, Bergheim
  - Boehringer Ingelheim, Bergisch Gladbach
  - Boehringer Ingelheim, Berkheim
  - Boehringer Ingelheim, Berlin
  - Boehringer Ingelheim, Berne
  - Boehringer Ingelheim, Bernsdorf
  - Boehringer Ingelheim, Betzdorf
  - Boehringer Ingelheim, Biebertal
  - Boehringer Ingelheim, Bielefeld
  - Boehringer Ingelheim, Bienenbüttel
  - Boehringer Ingelheim, Bippen
  - Boehringer Ingelheim, Birkenfeld
  - Boehringer Ingelheim, Birkenwerder
  - Boehringer Ingelheim, Blankenhain
  - Boehringer Ingelheim, Blaustein
  - Boehringer Ingelheim, Blieskastel
  - Boehringer Ingelheim, Bobritzsch
  - Boehringer Ingelheim, Bocholt
  - Boehringer Ingelheim, Bochum
  - Boehringer Ingelheim, Bockenem
  - Boehringer Ingelheim, Bodelshausen
  - Boehringer Ingelheim, Bodenfelde
  - Boehringer Ingelheim, Bodenkirchen
  - Boehringer Ingelheim, Bodenwöhr
  - Boehringer Ingelheim, Bodman-Ludwigshafen
  - Boehringer Ingelheim, Bollendorf
  - Boehringer Ingelheim, Bonn
  - Boehringer Ingelheim, Bopfingen
  - Boehringer Ingelheim, Borgholzhausen
  - Boehringer Ingelheim, Borken
  - Boehringer Ingelheim, Borna
  - Boehringer Ingelheim, Bornheim
  - Boehringer Ingelheim, Bottendorf
  - Boehringer Ingelheim, Bottmersdorf
  - Boehringer Ingelheim, Bottrop
  - Boehringer Ingelheim, Bovenden
  - Boehringer Ingelheim, Böhlen
  - Boehringer Ingelheim, Bösel
  - Boehringer Ingelheim, Brake
  - Boehringer Ingelheim, Brandenburg
  - Boehringer Ingelheim, Brannenburg
  - Boehringer Ingelheim, Braunschweig
  - Boehringer Ingelheim, Brechen
  - Boehringer Ingelheim, Breitenbrunn
  - Boehringer Ingelheim, Bremen
  - Boehringer Ingelheim, Bremerhaven
  - Boehringer Ingelheim, Brensbach
  - Boehringer Ingelheim, Breuberg
  - Boehringer Ingelheim, Bruchköbel
  - Boehringer Ingelheim, Brunsbüttel
  - Boehringer Ingelheim, Buchbach
  - Boehringer Ingelheim, Buckow
  - Boehringer Ingelheim, Buedelsdorf
  - Boehringer Ingelheim, Burg
  - Boehringer Ingelheim, Burgau
  - Boehringer Ingelheim, Burgdorf, Hanover
  - Boehringer Ingelheim, Burgpreppach
  - Boehringer Ingelheim, Burtenbach
  - Boehringer Ingelheim, Buttstädt
  - Boehringer Ingelheim, Butzbach
  - Boehringer Ingelheim, Bückeburg
  - Boehringer Ingelheim, Bünde
  - Boehringer Ingelheim, Büttelborn
  - Boehringer Ingelheim, Cadolzburg
  - Boehringer Ingelheim, Calbe
  - Boehringer Ingelheim, Calberlah
  - Boehringer Ingelheim, Castrop-Rauxel
  - Boehringer Ingelheim, Celle
  - Boehringer Ingelheim, Chemnitz
  - Boehringer Ingelheim, Cochem
  - Boehringer Ingelheim, Coppenbrügge
  - Boehringer Ingelheim, Crimmitschau
  - Boehringer Ingelheim, Crivitz
  - Boehringer Ingelheim, Cuxhaven
  - Boehringer Ingelheim, Dabel
  - Boehringer Ingelheim, Darmstadt
  - Boehringer Ingelheim, Dassow
  - Boehringer Ingelheim, Datteln
  - Boehringer Ingelheim, Daun
  - Boehringer Ingelheim, Deggendorf
  - Boehringer Ingelheim, Deidesheim
  - Boehringer Ingelheim, Deining
  - Boehringer Ingelheim, Delitzsch
  - Boehringer Ingelheim, Demen
  - Boehringer Ingelheim, Denkendorf
  - Boehringer Ingelheim, Dessau
  - Boehringer Ingelheim, Detmold
  - Boehringer Ingelheim, Dettenheim
  - Boehringer Ingelheim, Deuben
  - Boehringer Ingelheim, Deutzen
  - Boehringer Ingelheim, Diepholz
  - Boehringer Ingelheim, Dillingen
  - Boehringer Ingelheim, Dingolfing
  - Boehringer Ingelheim, Dinkelsbühl
  - Boehringer Ingelheim, Dinslaken
  - Boehringer Ingelheim, Dissen
  - Boehringer Ingelheim, Dogern
  - Boehringer Ingelheim, Dollern
  - Boehringer Ingelheim, Donaueschingen
  - Boehringer Ingelheim, Dormagen
  - Boehringer Ingelheim, Dornstetten
  - Boehringer Ingelheim, Dorsten
  - Boehringer Ingelheim, Dortmund
  - Boehringer Ingelheim, Dörentrup
  - Boehringer Ingelheim, Dörpen
  - Boehringer Ingelheim, Dreieich
  - Boehringer Ingelheim, Drensteinfurt
  - Boehringer Ingelheim, Dresden
  - Boehringer Ingelheim, Driedorf
  - Boehringer Ingelheim, Duderstadt
  - Boehringer Ingelheim, Duisburg
  - Boehringer Ingelheim, Dummerstorf
  - Boehringer Ingelheim, Düren
  - Boehringer Ingelheim, Düsseldorf
  - Boehringer Ingelheim, Ebergötzen
  - Boehringer Ingelheim, Ebermannstadt
  - Boehringer Ingelheim, Eberstadt
  - Boehringer Ingelheim, Ebhausen
  - Boehringer Ingelheim, Edewecht
  - Boehringer Ingelheim, Edling
  - Boehringer Ingelheim, Egelsbach
  - Boehringer Ingelheim, Ehingen
  - Boehringer Ingelheim, Eilenburg
  - Boehringer Ingelheim, Eisenhüttenstadt
  - Boehringer Ingelheim, Eiterfeld
  - Boehringer Ingelheim, Eitorf
  - Boehringer Ingelheim, Ellwangen
  - Boehringer Ingelheim, Elmshorn
  - Boehringer Ingelheim, Emersacker
  - Boehringer Ingelheim, Emmendingen
  - Boehringer Ingelheim, Emsdetten
  - Boehringer Ingelheim, Enger
  - Boehringer Ingelheim, Enkenbach-Alsenborn
  - Boehringer Ingelheim, Ennepetal
  - Boehringer Ingelheim, Ennigerloh
  - Boehringer Ingelheim, Eppstein
  - Boehringer Ingelheim, Erding
  - Boehringer Ingelheim, Erftstadt
  - Boehringer Ingelheim, Erkrath
  - Boehringer Ingelheim, Erligheim
  - Boehringer Ingelheim, Erndtebrück
  - Boehringer Ingelheim, Erolzheim
  - Boehringer Ingelheim, Eschborn
  - Boehringer Ingelheim, Eschelbronn
  - Boehringer Ingelheim, Eschweiler
  - Boehringer Ingelheim, Eslohe
  - Boehringer Ingelheim, Espenhain
  - Boehringer Ingelheim, Essen
  - Boehringer Ingelheim, Esslingen am Neckar
  - Boehringer Ingelheim, Euskirchen
  - Boehringer Ingelheim, Filderstadt
  - Boehringer Ingelheim, Floh-Seligenthal
  - Boehringer Ingelheim, Flöha
  - Boehringer Ingelheim, Forbach
  - Boehringer Ingelheim, Forchheim
  - Boehringer Ingelheim, Frankenberg
  - Boehringer Ingelheim, Frankenthal
  - Boehringer Ingelheim, Frankfurt
  - Boehringer Ingelheim, Freiberg
  - Boehringer Ingelheim, Freiburg im Breisgau
  - Boehringer Ingelheim, Freigericht
  - Boehringer Ingelheim, Freudenstadt
  - Boehringer Ingelheim, Freyung
  - Boehringer Ingelheim, Friedland
  - Boehringer Ingelheim, Friedrichshafen
  - Boehringer Ingelheim, Friedrichsthal
  - Boehringer Ingelheim, Frohburg
  - Boehringer Ingelheim, Fulda
  - Boehringer Ingelheim, Furtwangen im Schwarzwald
  - Boehringer Ingelheim, Fürstenwalde
  - Boehringer Ingelheim, Füssen
  - Boehringer Ingelheim, Gangelt
  - Boehringer Ingelheim, Gardelegen
  - Boehringer Ingelheim, Garmisch-Partenkirchen
  - Boehringer Ingelheim, Gars
  - Boehringer Ingelheim, Gebesee
  - Boehringer Ingelheim, Geesthacht
  - Boehringer Ingelheim, Gelbensande
  - Boehringer Ingelheim, Gelsenkirchen
  - Boehringer Ingelheim, Gensingen
  - Boehringer Ingelheim, Georgsmarienhütte
  - Boehringer Ingelheim, Gera
  - Boehringer Ingelheim, Gerbstedt
  - Boehringer Ingelheim, Germering
  - Boehringer Ingelheim, Germersheim
  - Boehringer Ingelheim, Gevelsberg
  - Boehringer Ingelheim, Giessen
  - Boehringer Ingelheim, Gifhorn
  - Boehringer Ingelheim, Gilserberg
  - Boehringer Ingelheim, Gladbeck
  - Boehringer Ingelheim, Gleichen
  - Boehringer Ingelheim, Goch
  - Boehringer Ingelheim, Gochsheim
  - Boehringer Ingelheim, Gomaringen
  - Boehringer Ingelheim, Göllheim
  - Boehringer Ingelheim, Göllingen
  - Boehringer Ingelheim, Göttingen
  - Boehringer Ingelheim, Grafenau
  - Boehringer Ingelheim, Gransee
  - Boehringer Ingelheim, Grassau
  - Boehringer Ingelheim, Greiz
  - Boehringer Ingelheim, Greven
  - Boehringer Ingelheim, Grevesmühlen
  - Boehringer Ingelheim, Griesheim
  - Boehringer Ingelheim, Gronau
  - Boehringer Ingelheim, Groß Grönau
  - Boehringer Ingelheim, Groß Quenstedt
  - Boehringer Ingelheim, Groß-Zimmern
  - Boehringer Ingelheim, Großalmerode
  - Boehringer Ingelheim, Großbottwar
  - Boehringer Ingelheim, Großefehn
  - Boehringer Ingelheim, Großhabersdorf
  - Boehringer Ingelheim, Großkorbetha
  - Boehringer Ingelheim, Großlangheim
  - Boehringer Ingelheim, Grömitz
  - Boehringer Ingelheim, Grünbach
  - Boehringer Ingelheim, Gummersbach
  - Boehringer Ingelheim, Güstrow
  - Boehringer Ingelheim, Haag
  - Boehringer Ingelheim, Hagen
  - Boehringer Ingelheim, Haigerloch
  - Boehringer Ingelheim, Haldensleben I
  - Boehringer Ingelheim, Halle
  - Boehringer Ingelheim, Hamburg
  - Boehringer Ingelheim, Hamm
  - Boehringer Ingelheim, Hamminkeln
  - Boehringer Ingelheim, Hanau
  - Boehringer Ingelheim, Hanerau-Hademarschen
  - Boehringer Ingelheim, Hanover
  - Boehringer Ingelheim, Harpstedt
  - Boehringer Ingelheim, Harsefeld
  - Boehringer Ingelheim, Harsewinkel
  - Boehringer Ingelheim, Haselünne
  - Boehringer Ingelheim, Hattersheim
  - Boehringer Ingelheim, Hattingen
  - Boehringer Ingelheim, Havixbeck
  - Boehringer Ingelheim, Hedersleben
  - Boehringer Ingelheim, Heek
  - Boehringer Ingelheim, Heide
  - Boehringer Ingelheim, Heidelberg
  - Boehringer Ingelheim, Heilbronn
  - Boehringer Ingelheim, Heimsheim
  - Boehringer Ingelheim, Heinsberg
  - Boehringer Ingelheim, Hellenthal
  - Boehringer Ingelheim, Hermaringen
  - Boehringer Ingelheim, Huska